CLINICAL TRIAL: NCT03409601
Title: The Role of Satiety in the Effect of Portion Size on Intake
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Additional outcome measures have been developed and added to the protocol.
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Barbara J. Rolls, BJR, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PortionSize104
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Feeding Behavior
Keywords: Obesity, eating behavior, food, nutrition
MeSH Terms: conditions — Feeding Behavior; Obesity | interventions — Portion Size

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 100% Portion Size (Experimental): Test meal consists of baseline (100%) portion size of meal.
  Interventions: Other: 100% Portion Size
- 125% Portion Size (Experimental): Test meal consists of food portion size that is 125% the size of baseline portion.
  Interventions: Other: 125% Portion Size
- 150% Portion Size (Experimental): Test meal consists of food portion size that is 150% the size of baseline portion.
  Interventions: Other: 150% Portion Size
- 175% Portion Size (Experimental): Test meal consists of food portion size that is 175% the size of baseline portion.
  Interventions: Other: 175% Portion Size

INTERVENTIONS:
Other: 100% Portion Size — Meal portion size at baseline
  Arms: 100% Portion Size
Other: 125% Portion Size — Meal portion size 125% of baseline
  Arms: 125% Portion Size
Other: 150% Portion Size — Meal portion size 150% of baseline
  Arms: 150% Portion Size
Other: 175% Portion Size — Meal portion size 175% of baseline
  Arms: 175% Portion Size

SUMMARY:
The study uses a crossover design in which the portion size of food is varied at each meal. Across four test meals, subjects will be served four different portions of food, and intake will be determined from pre- and post-meal food weights. The first visit will be a screening visit, at which subjects will complete the consent form, have their height and weight measured, and rate the taste of the study food. Test meals will be scheduled once a week for four weeks. At visits 2-5, subjects will eat lunch and rate characteristics of the meal. At visit 6, subjects will complete various questionnaires. The objective of this study is to determine whether any individual characteristics related to satiety influence the effect of portion size on intake.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to travel to Penn State University Park campus weekly for meals
* Be a man or woman 18 - 60 years old
* Regularly eat 3 meals/day
* Be willing to avoid alcohol the day before and during test days
* Have a body mass index between 18.0 and 35.0 kg/m-squared
* Be willing to refrain from eating after 10 pm the evening before test sessions

Exclusion Criteria:

* A smoker
* An athlete in training
* Pregnant or breastfeeding at the time of screening
* Have taken prescription or non-prescription drugs that may affect appetite or food intake within the last 3 months
* Dislike or be unable to eat the test foods (because of allergies, intolerance, or dietary restrictions)
* Currently dieting to gain or lose weight
* Have a health condition that affects appetite
* Have participated in a similar study in our lab in the past year

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Differences in energy intake | Weeks 1, 2, 3, and 4
  Calculated energy intake (kcal) based on weight and energy density of food consumed
Differences in intake by weight | Weeks 1, 2, 3, and 4
  Weights (grams) of all foods consumed

SECONDARY OUTCOMES:
Sensory-specific satiety | Weeks 1, 2, 3, and 4
  Change in taste pleasantness of eaten foods compared to uneaten foods
Eating rate | Weeks 1, 2, 3, and 4
  Assessed from meal duration and number of bites taken
Ratings of hunger and satiety | Weeks 1, 2, 3, and 4
  100-point visual analog scales
Ratings of sensory characteristics of the food | Weeks 1, 2, 3, and 4
  100-point visual analog scales
Ratings of meal characteristics | Weeks 1, 2, 3, and 4
  100-point visual analog scales

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No